CLINICAL TRIAL: NCT04897464
Title: Validation Study of a New Digital Treatment Test Based on Interactive Video Games for Alzheimer's Disease
Brief Title: Validation Study of a New Digital Treatment Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Braingaze (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT-AD-01
Record Dates: First submitted 2021-05-13; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Alzheimer Disease; MCI
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Other: BGaze therapy Alzheimer

INTERVENTIONS:
Other: BGaze therapy Alzheimer — BGaze Therapy is an interactive eye tracking game

SUMMARY:
Oculomotor behavior and cognitive processing of visual information are intimately connected. AD patients show ocular movement problems. Oculomotor deficits are broad consisting mainly of different saccade metrics, altered pupil responses. and smaller and irregular eye vergence movements. Here we test an interactive eye-tracking game to improve eye motion control and thereby training cognitive behavior

ELIGIBILITY:
Inclusion Criteria:

1) Clinical diagnosis of MCI or AD

Exclusion Criteria:

1. Severe cognitive deterioration
2. History of neurological disease with clinically relevant impact on cognition
3. Severe psychiatric disorder
4. Incidental structural brain findings with impact on cognitive impairment
5. Presence of relevant visual problems

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
MoCA | immediately after the intervention
  Measure changes in MoCA
MMSE | immediately after the intervention
  Measure changes in MMSE

SECONDARY OUTCOMES:
CANTAB | immediately after the intervention
  Measure changes in CANTAB tests

CONTACTS AND LOCATIONS:
Locations (1):
- Braingaze, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
anonymized data can be shared upon request